CLINICAL TRIAL: NCT02534870
Title: Multiple-Dose Pharmacokinetics, Safety and Tolerability of the Co-administration of ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) and ABT-333 in Healthy Chinese Subjects
Brief Title: Pharmacokinetics and Safety of the Co-administration of ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) and ABT-333 in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-769
Record Dates: First submitted 2015-08-26; First posted 2015-08-28 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Healthy Volunteer
Keywords: Volunteer
MeSH Terms: interventions — paritaprevir; dasabuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-450/r/ABT-267 + ABT-333 (Experimental): ABT-450/r/ABT-267 will be administered once daily in the morning and ABT-333 will be administered in the morning and evening for 14 days.
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333

INTERVENTIONS:
Drug: ABT-450/r/ABT-267 — Tablet
  Other Names: Paritaprevir/Ritonavir/Ombitasvir
Drug: ABT-333 — Tablet
  Other Names: Dasabuvir

SUMMARY:
The purpose of this study is to assess the pharmacokinetics and safety of multiple oral doses of ABT-450/ritonavir/ABT-267 and ABT-333 when co-administered under non-fasting conditions in healthy Chinese adult participants.

ELIGIBILITY:
Inclusion Criteria: Participant must be Chinese (i.e., of Chinese ancestry).

If female, participant must be either postmenopausal for at least 2 years, surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or practicing at least one of the following methods of birth control with male partner(s): total abstinence from sexual intercourse as the preferred life style of the subject, periodic abstinence is not acceptable; vasectomized partner(s); hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration; intrauterine device (IUD); or double-barrier method (condoms, contraceptive sponge, or diaphragm with spermicidal jellies or creams)

Hormonal contraceptives, including but not limited to oral, topical, injectable or implantable varieties, may not be used during the study.

If male, the participant must be surgically sterile or practicing at least 1 of the following methods of contraception, and refrain from sperm donation, from initial study drug administration until 90 days after the last dose of study drug: partner(s) using an IUD; partner(s) using oral, injected, intravaginal, or implanted methods of hormonal contraceptives; participant and/or partner(s) using double-barrier method (condoms, contraceptive sponge, diaphragm with spermicidal jellies or creams, or vaginal ring); or total abstinence from sexual intercourse as the preferred life style of the subject; periodic abstinence is not acceptable

Body Mass Index (BMI) is ≥ 18 to < 30 kg/m^2.

A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, a 12-lead electrocardiogram (ECG) and chest x-ray (CXR).

Exclusion Criteria: Use of any medications (prescription and over-the-counter), vitamins and/or herbal supplements within the 2-week period prior to the first dose of study drug administration or within 10 half-lives of the respective medication, whichever is longer.

History of epilepsy, any clinically significant cardiovascular, respiratory (except mild asthma), renal, hepatic, gastrointestinal, hematologic, neurologic, thyroid, or any uncontrolled medical illness or psychiatric disease or disorder.

Clinically significant abnormal ECG: ECG with QT interval corrected for heart rate using Fridericia's correction formula (QTcF) > 450 msec in females and > 430 msec in males, or ECG with second or third degree atrioventricular block.

Previous exposure to more than a single dose of ABT-450/r/ABT-267, or ABT-333 within the past 12 weeks, or previous participation in this study.

Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive ABT-450, ritonavir, ABT-267, or ABT-333.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of ABT-450 | Prior to the morning dose (0 hour) and 1, 2, 3, 4, 6, 9, 12, 15, 18, and 24 hours after the morning dose on Study Days 1 and 14; and 36, 48, and 72 hours after the morning dose on Study Day 14
  Cmax is the highest concentration that a drug achieves in the blood after administration in a dosing interval.
Maximum Plasma Concentration (Cmax) of ABT-267 | Prior to the morning dose (0 hour) and 1, 2, 3, 4, 6, 9, 12, 15, 18, and 24 hours after the morning dose on Study Days 1 and 14; and 36, 48, and 72 hours after the morning dose on Study Day 14
  Cmax is the highest concentration that a drug achieves in the blood after administration in a dosing interval.
Maximum Plasma Concentration (Cmax) of ABT-333 | Prior to the morning dose (0 hour) and 1, 2, 3, 4, 6, 9, 12, 15, 18, and 24 hours after the morning dose on Study Days 1 and 14; and 36, 48, and 72 hours after the morning dose on Study Day 14
  Cmax is the highest concentration that a drug achieves in the blood after administration in a dosing interval.
Maximum Plasma Concentration (Cmax) of Ritonavir | Prior to the morning dose (0 hour) and 1, 2, 3, 4, 6, 9, 12, 15, 18, and 24 hours after the morning dose on Study Days 1 and 14; and 36, 48, and 72 hours after the morning dose on Study Day 14
  Cmax is the highest concentration that a drug achieves in the blood after administration in a dosing interval.
Time to Maximum Plasma Concentration (Tmax) of ABT-450 | Prior to the morning dose (0 hour) and 1, 2, 3, 4, 6, 9, 12, 15, 18, and 24 hours after the morning dose on Study Days 1 and 14; and 36, 48, and 72 hours after the morning dose on Study Day 14
  Tmax is the time it takes for a drug to achieve Cmax.
Time to Maximum Plasma Concentration (Tmax) of ABT-267 | Prior to the morning dose (0 hour) and 1, 2, 3, 4, 6, 9, 12, 15, 18, and 24 hours after the morning dose on Study Days 1 and 14; and 36, 48, and 72 hours after the morning dose on Study Day 14
  Tmax is the time it takes for a drug to achieve Cmax.
Time to Maximum Plasma Concentration (Tmax) of ABT-333 | Prior to the morning dose (0 hour) and 1, 2, 3, 4, 6, 9, 12, 15, 18, and 24 hours after the morning dose on Study Days 1 and 14; and 36, 48, and 72 hours after the morning dose on Study Day 14
  Tmax is the time it takes for a drug to achieve Cmax.
Time to Maximum Plasma Concentration (Tmax) of Ritonavir | Prior to the morning dose (0 hour) and 1, 2, 3, 4, 6, 9, 12, 15, 18, and 24 hours after the morning dose on Study Days 1 and 14; and 36, 48, and 72 hours after the morning dose on Study Day 14
  Tmax is the time it takes for a drug to achieve Cmax.
Trough Concentration (Ctrough) of ABT-450 | Prior to the morning dose on Study Days 7, 9, 11, 13 and 14; 24 hours after Day 14 dose
  Ctrough is the lowest concentration of a drug in the blood after administration in a dosing interval.
Trough Concentration (Ctrough) of ABT-267 | Prior to the morning dose on Study Days 7, 9, 11, 13 and 14; 24 hours after Day 14 dose
  Ctrough is the lowest concentration of a drug in the blood after administration in a dosing interval.
Trough Concentration (Ctrough) of ABT-333 | Prior to the morning dose on Study Days 7, 9, 11, 13 and 14; 24 hours after Day 14 dose
  Ctrough is the lowest concentration of a drug in the blood after administration in a dosing interval.
Trough Concentration (Ctrough) of Ritonavir | Prior to the morning dose on Study Days 7, 9, 11, 13 and 14; 24 hours after Day 14 dose
  Ctrough is the lowest concentration of a drug in the blood after administration in a dosing interval.
Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC24) Post-dose of ABT-450 | Prior to the morning dose (0 hour) and 1, 2, 3, 4, 6, 9, 12, 15, 18, and 24 hours after the morning dose on Study Days 1 and 14
Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC24) Post-dose of Ritonavir | Prior to the morning dose (0 hour) and 1, 2, 3, 4, 6, 9, 12, 15, 18, and 24 hours after the morning dose on Study Days 1 and 14
Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC24) Post-dose of ABT-267 | Prior to the morning dose (0 hour) and 1, 2, 3, 4, 6, 9, 12, 15, 18, and 24 hours after the morning dose on Study Days 1 and 14
Area Under the Plasma Concentration-time Curve From 0 to 12 Hours (AUC12) Post-dose of ABT-333 | Prior to the morning dose (0 hour) and 1, 2, 3, 4, 6, 9, and 12 hours after the morning dose on Study Days 1 and 14
Number of participants with adverse events | Daily for approximately 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Yan Luo, MD, Study Director — AbbVie
Locations (1):
- Site Reference ID/Investigator# 137655, Shanghai, China

REFERENCES:
- [Derived] Zha J, Ding B, Wang H, Zhao W, Yu C, Alves K, Mobashery N, Luo Y, Menon RM. Pharmacokinetics of Ombitasvir, Paritaprevir, Ritonavir, and Dasabuvir in Healthy Chinese Subjects and HCV GT1b-Infected Chinese, South Korean and Taiwanese Patients. Eur J Drug Metab Pharmacokinet. 2019 Feb;44(1):43-52. doi: 10.1007/s13318-018-0492-8. PMID 29909549